CLINICAL TRIAL: NCT04084782
Title: An Internet Mediated Research Study to Assess the Quality of Life of Consumers With Self-reported Fungal Nail Infection (Onychomycosis) During Treatment With Scholl Fungal Nail.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: NPD89101
Record Dates: First submitted 2019-08-09; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Onychomycosis of Toenail
Keywords: Fungal Nail Infection; Internet Mediated Research Study
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Onychomycosis group: Subjects in this group suffer from onychomycosis of the toenail, who chose to self treat by purchasing the product from an online platform.
  Interventions: Device: Fungal Nail Treatment Kit

INTERVENTIONS:
Device: Fungal Nail Treatment Kit — The treatment kit consists of 5 disposable nail files to be used to remove the top layer of the infected nail at various times throughout the use of the product and a liquid formulation and brush applicator.

SUMMARY:
To evaluate the effect on quality of life of consumers with self-reported onychomycosis during the first 4 weeks of treatment in relation to the appearance of the infected toenail.

DETAILED DESCRIPTION:
The appearance of the infected toe nail in those suffering from the disease may have a greater impact on quality of life than the severity of the disease. It is believed that a visual improvement in the appearance of the infected toenail at an earlier stage could have a positive impact on quality of life and encourage compliance with treatment. The aim of this consumer study is to evaluate the quality of life of consumers with onychomycosis and investigate its relation to the appearance of the infected toenail within the initial 4 weeks of treatment with Scholl Fungal Nail following its purchase from an eCommerce platform.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Consumers who have purchased the product online
* Consumers who are willing to participate in the study

Exclusion Criteria:

* Female consumers who are pregnant or breast feeding
* Participants with Diabetes (Type I or II)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is targeting consumers who chose to self-treat by purchasing the Fungal Nail product from the eCommerce platform. Only consumers who agree to participate in the consumer study after reviewing the information provided and provide electronic Consent will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-08-13 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Improvement | 28 days
  Change in mean total score of the OnyCOE-t™ from baseline to end of inital treatment period. The domains are transformed into 0-100 scale where higher scores indicate better functioning. Changes from baseline of the mean total score will be evaluated with repeated measures t-tests.
  The questionnaire contains 7 domains:
  7-item Toenail Symptoms, containing Symptom Frequency (5 categories: 1 = never, 5 = very often) and Symptom Bothersomeness (5 categories: 1 = not at all bothered, 5 = extremely bothered) 8-item Appearance Problems (4 categories: 1 = very much a problem, 4 = not a problem) 7-item Physical Activities Problems (4 categories: 1 = very much a problem, 4 = not a problem)
  1-item Overall Problem (4 categories; 1 = very much a problem, 4 = not a problem) 7-item Stigma (5 categories: 0 = does not describe me at all, 4 = describes me very well) 3-item Treatment Satisfaction scale (5 categories: 1 = very satisfied, 5 very dissatisfied)

SECONDARY OUTCOMES:
Participant perception of the improvement in healthy appearance of their infected toenail. | Any timepoint up to day 28
  The participants will be asked to score the statement "My toenail looks healthy" (prior to product use) and "My toenail looks healthier" (at various time points following product application) using the following categories, strongly agree, agree, neither agree nor disagree, disagree, Strongly disagree. A successful outcome of this measure would be 70% Top 2 Boxes (T2B) (Strongly Agree or Agree) improvement in the healthier appearance of the target toenail at any post baseline assessment compare to Day 1 (prior to initial product application)
Participant perception of improvement in brightness of their infected toenail. | Any timepoint up to day 28
  The participants will be asked to score the statement "My toenail looks bright" (prior to product use) and "My toenail looks brighter" (at various time points following product application) using the following categories, strongly agree, agree, neither agree nor disagree, disagree, Strongly disagree. A successful outcome of this measure would be 70% T2B (Strongly Agree or Agree) improvement in the brighter appearance of the target toenail as determined by participant perceived questions at any post baseline assessment compare to Day 1 (prior to initial product application)
Participant perception of the improvement in colour of their infected toenail. | Any timepoint up to day 28
  The participants will be asked to score the statement "My toenail is its natural colour" (prior to product use) and "My toenail is returning to its natural colour" (at various time points following product application) using the following categories, strongly agree, agree, neither agree nor disagree, disagree, Strongly disagree. A successful outcome of this measure would be 70% T2B (Strongly Agree or Agree) improvement in the colour of the target toenail as determined by participant perceived questions at any post baseline assessment compare to Day 1 (prior to initial product application)
Participant perception of the improvement in smoothness of their infected toenail. | Any timepoint up to day 28
  The participants will be asked to score the statement "My toenail looks smooth" (prior to product use) and "My toenail looks smoother" (at various time points following product application) using the following categories, strongly agree, agree, neither agree nor disagree, disagree, Strongly disagree. A successful outcome of this measure would be 70% T2B (Strongly Agree or Agree) improvement in the smoothness of the target toenail as determined by participant perceived questions at any post baseline assessment compare to Day 1 (prior to initial product application)
Participant perception of improvement of their feelings of embarrassment associated with their infected toenail. | Any timepoint up to day 28
  The participants will be asked to score the statement "I am feeling embarrassed by the appearance of my toenail" (prior to product use and at various time points following product application) using the following categories, strongly agree, agree, neither agree nor disagree, disagree, Strongly disagree. A successful outcome of this measure would be 70% of responses show improvement from baseline and are in the T2B (Strongly Disagree or Disagree) in the feelings of embarrassment relating to the appearance of the target toenail as determined by participant perceived questions at any post baseline assessment compared to Day 1 (prior to initial product application)
Individual OnyCOE-t(TM) domain improvement | 28 days
  Improvement in the mean scores on the individual OnyCOE-t(TM) domains (as detailed in outcome 1 above).
  The data will be summarised with means, standard deviations, range and 95% confidence intervals, changes from baseline of the mean individual domain score will be evaluated using repeated measures t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Fawkes, MBChB, Principal Investigator — Reckitt Bencksier, Dansom Lane, Hull
Locations (1):
- RB Health, Hull, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The study sponsor may author journal article outlining the collective results of the study, however IPD will not be shared.

REFERENCES:
- [Background] Velasquez-Agudelo V, Cardona-Arias JA. Meta-analysis of the utility of culture, biopsy, and direct KOH examination for the diagnosis of onychomycosis. BMC Infect Dis. 2017 Feb 22;17(1):166. doi: 10.1186/s12879-017-2258-3. PMID 28222676
- [Background] Sigurgeirsson B, Ghannoum MA, Osman-Ponchet H, Kerrouche N, Sidou F. Application of cosmetic nail varnish does not affect the antifungal efficacy of amorolfine 5% nail lacquer in the treatment of distal subungual toenail onychomycosis: results of a randomised active-controlled study and in vitro assays. Mycoses. 2016 May;59(5):319-26. doi: 10.1111/myc.12473. Epub 2016 Feb 11. PMID 26867498
- [Background] Christenson JK, Peterson GM, Naunton M, Bushell M, Kosari S, Baby KE, Thomas J. Challenges and Opportunities in the Management of Onychomycosis. J Fungi (Basel). 2018 Jul 24;4(3):87. doi: 10.3390/jof4030087. PMID 30042327
- [Background] Tosti A, Elewski BE. Treatment of onychomycosis with efinaconazole 10% topical solution and quality of life. J Clin Aesthet Dermatol. 2014 Nov;7(11):25-30. PMID 25489379
- [Background] Potter LP, Mathias SD, Raut M, Kianifard F, Tavakkol A. The OnyCOE-t questionnaire: responsiveness and clinical meaningfulness of a patient-reported outcomes questionnaire for toenail onychomycosis. Health Qual Life Outcomes. 2006 Aug 15;4:50. doi: 10.1186/1477-7525-4-50. PMID 16911778
- [Background] Potter LP, Mathias SD, Raut M, Kianifard F, Landsman A, Tavakkol A. The impact of aggressive debridement used as an adjunct therapy with terbinafine on perceptions of patients undergoing treatment for toenail onychomycosis. J Dermatolog Treat. 2007;18(1):46-52. doi: 10.1080/09546630600965004. PMID 17373090
- See also: UK Research Integrity Office - Good Practice in research: internet mediated research V1.0 Dec 2016 — https://ukrio.org/wp-content/uploads/UKRIO-Guidance-Note-Internet-Mediated-Research-v1.0.pdf